CLINICAL TRIAL: NCT05732922
Title: Optimising Remote Consulting and Home Assessment of Medically Vulnerable Rural Patients During Unscheduled and Planned Primary Care- Assessing Feasibility of the ORCHARD Intervention
Brief Title: ORCHARD- Optimising Home Assessment of Rural Patients
Acronym: ORCHARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 310499
Record Dates: First submitted 2022-10-25; First posted 2023-02-17 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Organ Transplant; Cancer; Inborn Errors of Metabolism; Immunosuppression; COPD Asthma; Sickle Cell Disease
Keywords: telemedicine; rurality; diagnostic equipment; vulnerable patients
MeSH Terms: conditions — Neoplasms; Metabolism, Inborn Errors; Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will be receiving their standard medical care.
- Intervention (Active Comparator): Participants will be receiving the intervention on top of their standard medical care.
  Interventions: Device: A sphygmanometer, a digital thermometer, a pulse oximeter and a peak flow meter will be given to participants to use during their telemedicine consultations with health care providers.

INTERVENTIONS:
Device: A sphygmanometer, a digital thermometer, a pulse oximeter and a peak flow meter will be given to participants to use during their telemedicine consultations with health care providers. — A sphygmanometer, a digital thermometer, a pulse oximeter and a peak flow meter will be given to participants in the intervention arm to use during their telemedicine consultations with health care providers.
  Arms: Intervention

SUMMARY:
This project assesses feasibility of providing medically vulnerable rural patients with Medical-Self-Assessment-Boxes containing equipment to use at home during telephone and video consultations (telemedicine) with GPs and other healthcare professionals. COVID-19 has caused an upsurge in primary care telemedicine which the investigators believe can be sustained and optimized to make things better for medically vulnerable rural patients beyond the pandemic. The investigators will achieve this by equipping the participants to self-measure and report key clinical measurements (e.g. blood pressure, temperature, oxygen levels) during telemedicine consultations. Before conducting a major evaluation of the Medical-Self-Assessment-Box for medically vulnerable rural patients the investigators must establish three things: First, to show the investigators can issue a Medical-Self-Assessment-Box to medically vulnerable rural patients and enable them to use it properly. Second, to determine that patients can use the Medical-Self-Assessment-Box effectively during telemedicine consultations. Third, to show that it is possible to measure how well the Medical-Self-Assessment-Box is working by counting how often the boxes are being used and whether use is appropriate and helpful. The knowledge gained will provide the investigators with the information needed to develop a funding proposal to evaluate Medical-Self-Assessment-Boxes for medically vulnerable rural patients in the whole of the UK.

ELIGIBILITY:
Inclusion Criteria:

* ● Solid organ transplant recipient

  * On the COVID-19 shielding list
  * People with specific cancers

    * People with cancer who had chemotherapy within the last 2 years
    * People with lung cancer that have had radical radiotherapy within the last two years
    * People with cancer of the blood or bone marrow such as leukaemia, lymphoma or myeloma who are at end stage treatment
    * People that have had immunotherapy or other continuing antibody treatments for cancer within the last two years
    * People that had other targeted cancer treatment which can affect the immune system, such as protein kinase inhibitors or PARP inhibitors within the last two years
    * People who had bone marrow or stem cell transplants in the last 6 months, or who are still taking immunosuppression drugs
  * People with severe respiratory conditions including all cystic fibrosis, severe asthma, and severe COPD
  * People with rare diseases and inborn errors of metabolism that significantly increase the risk of infections (such as SCID, homozygous sickle cell anaemia)
  * People in immunosuppression therapies sufficient to significantly increase risk of infection

Inclusion criteria for GPs:

* A GP working at the pilot study practice and carried out telemedicine consultations with participants
* A GP who can provide informed consent

Exclusion Criteria:

* People whose GP feels they are not able to participate in the research. People unable to consent to participate. Non-English speakers

Exclusion criteria for GPs:

A GP that cannot provide informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Short questionnaire | 6 months (given at the end of every TM consultation)
  The questionnaire will assess use of equipment, perception of how helpful the equipment was for the consultation and the reasons why it was helpful.
Interviews | 1 day (end of study interview)
  Qualitative data collected at the end of the study according to a topic guide.

SECONDARY OUTCOMES:
Number of consultations face to face | 6 months (every time there is a consultation)
  Number of face to face consultations
Number of consultations TM | 6 months (every time there is a consultation)
  Number of telemedicine consultations
Hospital admissions elective | 6 months (every time there is an admission)
  Number of elective hospital admissions
Hospital admissions emergency | 6 months (every time there is an admission)
  Number of emergency hospital admissions
Ambulance service call-outs | 6 months (every time there is a call-out)
  Number of Scottish ambulance service call-outs
Ambulance service paramedics | 6 months (every time there is an assessment)
  Number of face-to-face paramedic assessment
Survival | 6 months (assessed at the end of the study)
  Survival at six months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Murchie, Principal Investigator — University of Aberdeen
Locations (1):
- University of Aberdeen, Aberdeen, Aberdeen City, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided